CLINICAL TRIAL: NCT00577629
Title: Dose-Intensive Chemotherapy Combined With Monoclonal Antibody Therapy and Targeted Radioimmunotherapy for Untreated Patients With High-Risk B-Cell Non-Hodgkin's Lymphoma
Brief Title: Chemotherapy With Monoclonal Antibody and Radioimmunotherapy for High-Risk B-Cell Non-Hodgkins Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00007096; GSK-103421 (Other Grant/Funding Number: GSK); 5762 (Other: DUMC old IRB #)
Record Dates: First submitted 2007-12-18; First posted 2007-12-20 (Estimated); Results first posted 2013-04-15 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Lymphoma, B-Cell
Keywords: high risk non-hodgkins lymphoma; NHL; Bexxar; high dose chemotherapy
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — Cyclophosphamide; Etoposide; Rituximab; Cytarabine; Doxorubicin; tositumomab I-131

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Induction + Consolidation + Bexxar (Experimental): Induction:Cyclophosphamide, Etoposide, and Rituxan (rituximab) followed by Consolidation: Cytarabine and Doxorubicin followed by radioimmunotherapy: Bexxar (tositumomab)
  Interventions: Drug: cyclophosphamide; Drug: etoposide; Drug: rituximab; Drug: cytarabine; Drug: doxorubicin; Drug: tositumomab

INTERVENTIONS:
Drug: cyclophosphamide — 1.5g/m2 IV over 1 hour on days 1-4 of induction for a total dose of 6.0g/m2
  Other Names: Cytoxan®
Drug: etoposide — 300mg/m2 IV over 1 hour every 12 on days 1-3 of induction for a total dose of 1.8 g/m2.
  Other Names: VP-16
Drug: rituximab — 375mg/m2 each week x 4 weeks of induction, beginning on day 1
  Other Names: Rituxan
Drug: cytarabine — 3g/m2 IV over 1 hour every 12 during consolidation for a total of 8 doses
  Other Names: Ara-C
Drug: doxorubicin — 45mg/m2/day IV over 30 minutes on days 1, 2, 3 during consolidation
  Other Names: Adriamycin
Drug: tositumomab — 450mg unlabeled tositumomab over 1 hour, followed by 5 millicurie (mCi) Iodine I-131 labeled tositumomab over 20 minutes on day 0. Therapeutic dose of labeled tositumomab will be administered on day 15.
  Other Names: Bexxar

SUMMARY:
The purpose of this study is to determine whether using high-dose chemotherapy, monoclonal antibodies, and targeted radioimmunotherapy will slow the progression of disease in patients with high-risk Non-Hodgkin's Lymphoma (NHL).

DETAILED DESCRIPTION:
This is a phase II efficacy trial for patients with untreated, high-risk, B-cell Non-Hodgkin's Lymphoma. The study will evaluate the efficacy and safety of high-dose chemotherapy combined with monoclonal antibodies and targeted radioimmunotherapy in previously untreated patients with high-risk NHL

ELIGIBILITY:
Inclusion Criteria:

* Untreated, biopsy proven B-cell non-Hodgkin's lymphoma
* Age >/= 18 years
* No other prior malignancy except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease-free for one year. The patient cannot have been exposed to chemotherapy to treat any of these diseases for at least 3 years prior to study entry.
* Meet staging studies and laboratory tests prior to induction, consolidation and radioimmunotherapy.

Exclusion Criteria:

* Significant medical and/or psychiatric illness which may compromise planned treatment;
* Pregnant or lactating;
* HIV-infection.
* Patients with follicular lymphoma grade 1, 2 or 3A are not eligible for this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2005-06-18 (Actual); Primary Completion 2012-04-08 (Actual); Study Completion 2016-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Rizzieri, MD, Principal Investigator — Duke Unversity Medical Center
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited between September 2005 and March 2011 at Duke University Medical Center.
Groups:
- All Subjects: Induction:Cyclophosphamide, Etoposide, and Rituxan followed by Consolidation:Cytarabine and Doxorubicin followed by radioimmunotherapy:Bexxar
Period: Treatment Period
Arm/Group | All Subjects
Started | 39
Completed | 38
Not Completed | 1
Not completed — Death | 1
Period: Long Term Follow-Up
Arm/Group | All Subjects
Started | 38
Completed | 13
Not Completed | 25
Not completed — Death | 15
Not completed — Lost to Follow-up | 5
Not completed — Withdrawal by Subject | 4
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Subjects
Number analyzed (Participants) | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 14
Age, Customized [Mean (Full Range); unit: Years] | 60 [21 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 27
Region of Enrollment [Number; unit: participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: 1 Year Progression-free Survival Rate
Description: Progression-free survival is measured from the first day of induction chemotherapy to the date of progression, relapse or death. Definitions of response criteria are as described by Cheson. Progressive Disease: >50% increase from nadir in the sum of the products of the greatest diameters (SPD) of any previously identified abnormal node for PDs or nonresponders, appearance of any new lesion during or at the end of therapy.
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Experimental: Induction + Consolidation + Bexxar: Induction: Cyclophosphamide, Etoposide, and Rituxan followed by Consolidation: Cytarabine and Doxorubicin followed by radioimmunotherapy: Bexxar
Arm/Group | Experimental: Induction + Consolidation + Bexxar
Number analyzed (Participants) | 39
percentage of participants | 0.74 [0.635 to 0.91]

2. Secondary Outcome: Disease-free Survival
Description: Disease-free survival is measured from the date of CR or CRu to date of relapse or death
Time Frame: 10 years
Population: Subjects who achieved a complete response. 9 patients experienced disease progression; 4 patients died.
  4 patients were lost-to-follow-up and 11 patients are still living, so DFS was calculated using the last date of follow-up.
Measure: Mean (Full Range); unit: months
Groups:
- Experimental: Induction + Consolidation + Bexxar: Induction:Cyclophosphamide, Etoposide, and Rituxan followed by Consolidation:Cytarabine and Doxorubicin followed by radioimmunotherapy: Bexxar
Arm/Group | Experimental: Induction + Consolidation + Bexxar
Number analyzed (Participants) | 29
months | 54.10 [2 to 116]

3. Secondary Outcome: Overall Survival
Description: Overall Survival is measured from the first day of chemotherapy until death from any cause.
Time Frame: 10 years
Population: All subjects who received chemotherapy
Measure: Number; unit: percentage of participants
Arm/Group | Experimental: Induction + Consolidation + Bexxar
Number analyzed (Participants) | 39
percentage of participants | 82

4. Secondary Outcome: Overall Response
Description: Percent of subjects who achieved a complete response (CR) or partial response (PR) any time during the treatment period.
  CR = complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present before therapy.
  PR =
  1. >/= 50% decrease in sum of the product of the diameters (SPD) of up to six of the largest dominant nodes or nodal masses.
  2. No increase should be observed in the size of other nodes, liver, or spleen.
  3. Splenic and hepatic nodules must regress by ≥ 50% in their SPD or, for single nodules, in the greatest transverse diameter.
  4. Except splenic and hepatic nodules, involvement of other organs is usually assessable and no measurable disease should be present.
  5. Patients who achieve a CR by the above criteria, but who have persistent morphologic bone marrow involvement will be considered partial responders.
  6. No new sites of disease should be observed.
Time Frame: up to 1 year
Measure: Number; unit: percentage of participants
Groups:
- Experimental: Induction + Consolidation + Bexxar: Induction: Cyclophosphamide, Etoposide, and Rituxan followed by Consolidation: Cytarabine and Doxorubicin followed by radioimmunotherapy: Bexxar)
Arm/Group | Experimental: Induction + Consolidation + Bexxar
Number analyzed (Participants) | 38
percentage of participants | 92

5. Secondary Outcome: Secondary Malignancies
Description: The number of patients who develop secondary malignancies including solid tumors, acute leukemia and myelodysplasia or other bone marrow failure syndromes.
Time Frame: 10 years
Population: All patients who received chemotherapy
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Induction + Consolidation + Bexxar
Number analyzed (Participants) | 39
Participants
  Myelodysplastic Syndrome (MDS) | 3
  Acute Myeloid Leukemia (AML) | 1
  Pancreatic Cancer | 1
  Hodgkins Lymphoma | 1
  Melanoma | 1
  Renal Cell Carcinoma | 1

ADVERSE EVENTS:
Time Frame: 2 years from the start of treatment with the following exception: data on malignancies/bone marrow failures will be collected for 10 years.
Description: All adverse events are reported whether or not they are considered related to study regimen.
Arm/Group | Experimental: Induction + Consolidation + Bexxar
Serious Adverse Events (participants affected / at risk) | 28/39
Other Adverse Events (participants affected / at risk) | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Induction + Consolidation + Bexxar (N=39)
Supraventricular and nodal arrhythmia - Atrial fibrillation (Cardiac disorders) | 1 (1)
Speech impairment (e.g., dysphasia or aphasia) (Nervous system disorders) | 1 (1)
Thrombosis / thrombus / embolism (Vascular disorders) | 1 (1)
Ataxia (incoordination) (Nervous system disorders) | 1 (1)
Thrombosis / embolism (vascular access-related) (Surgical and medical procedures) | 1 (1)
Gastrointestinal - Other (Gastrointestinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Dermatology / Skin - Other (Skin and subcutaneous tissue disorders) | 1 (1)
Leukocytes (total WBC) (Investigations) | 1 (1)
Cardiac Arrhythmia - Other (Cardiac disorders) | 1 (1)
Ascites (non-malignant) (Gastrointestinal disorders) | 1 (1)
Infection with unknown ANC - Lung (pneumonia) (Infections and infestations) | 1 (1)
Hemorrhage, pulmonary / upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 2 (2)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 2 (2)
Pain - Abdomen NOS (Gastrointestinal disorders) | 2 (2)
Mucositis / Stomatitis (clinical exam) (Gastrointestinal disorders) | 3 (3)
Febrile neutropenia (fever of unknown origin without documented infection) (Blood and lymphatic system disorders) | 4 (4)
Infection - Other (Infections and infestations) | 4 (5)
Malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (Infections and infestations) | 5 (6)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Induction + Consolidation + Bexxar (N=39)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Supraventricular and nodal arrhythmia - Atrial fibrillation (Cardiac disorders) | 2 (2)
Esophagitis (Gastrointestinal disorders) | 2 (2)
Hemorrhage, pulmonary / upper respiratory (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Edema (General disorders) | 2 (2)
Edema: Other (General disorders) | 2 (2)
Memory Impairment (Nervous system disorders) | 2 (2)
Neuropathy: motor (Nervous system disorders) | 2 (2)
Speech impairment (e.g., dysphasia or aphasia) (Nervous system disorders) | 2 (2)
Tremor (Nervous system disorders) | 2 (2)
Pain - Chest / thorax NOS (General disorders) | 2 (2)
Pain - Rectum (Gastrointestinal disorders) | 2 (2)
Pain - Sinus (Nervous system disorders) | 2 (2)
Pain-Pulmonary / Upper Respiratory (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pain-Renal / Genitourinary (Gastrointestinal disorders) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 2 (2)
Left ventricular systolic dysfunction (Cardiac disorders) | 3 (3)
Hemorrhage, GI (Gastrointestinal disorders) | 3 (3)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 3 (3)
Confusion (Psychiatric disorders) | 3 (3)
Mood Alteration - Agitation (Psychiatric disorders) | 3 (3)
Somnolence / depressed level of consciousness (Nervous system disorders) | 3 (3)
Pain (General disorders) | 3 (3)
Voice changes / dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Thrombosis / thrombus / embolism (Vascular disorders) | 3 (3)
Weight gain (Investigations) | 4 (4)
Dry mouth / salivary gland (xerostomia) (Gastrointestinal disorders) | 3 (4)
Hemorrhage, pulmonary / upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 4 (4)
Ataxia (incoordination) (Nervous system disorders) | 3 (4)
Psychosis (hallucinations / delusions) (Psychiatric disorders) | 4 (4)
Pain - Oral cavity (Gastrointestinal disorders) | 3 (4)
Palpitations (Cardiac disorders) | 5 (5)
Metabolic / Laboratory - Other (Investigations) | 3 (5)
Pain - Throat / pharynx / larynx (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Renal / Genitourinary - Other (Renal and urinary disorders) | 4 (5)
Supraventricular and nodal arrhythmia (Cardiac disorders) | 4 (6)
Hot flashes / flushes (Vascular disorders) | 5 (6)
Mucositis / stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 5 (6)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 6 (6)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 6 (6)
Vision - blurred vision (Eye disorders) | 6 (6)
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 5 (6)
Thrombosis / embolism (vascular access-related) (Surgical and medical procedures) | 5 (6)
Weight loss (Investigations) | 7 (7)
Pruritus / itching (Skin and subcutaneous tissue disorders) | 6 (7)
Pain - Abdomen NOS (Gastrointestinal disorders) | 5 (7)
Pain - Back (Musculoskeletal and connective tissue disorders) | 5 (7)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 8 (8)
Gastrointestinal - Other (Gastrointestinal disorders) | 7 (8)
Taste Alteration (dysgeusia) (Nervous system disorders) | 8 (8)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 6 (8)
Pain - Head / headache (Nervous system disorders) | 7 (8)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 6 (9)
Heartburn / dyspepsia (Gastrointestinal disorders) | 9 (9)
Mood Alteration - Anxiety (Psychiatric disorders) | 7 (9)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 6 (9)
Rigors / chills (General disorders) | 9 (10)
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 10 (10)
Infection - Other (Infections and infestations) | 9 (10)
Hypotension (Vascular disorders) | 9 (11)
Pain-Musculoskeletal (Musculoskeletal and connective tissue disorders) | 8 (11)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 11 (12)
Creatinine (Investigations) | 9 (12)
Dry Skin (Skin and subcutaneous tissue disorders) | 11 (13)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 12 (13)
Muscle weakness, generalized or specific area (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 12 (13)
Neurology - Other (Nervous system disorders) | 8 (13)
Joint-function (Musculoskeletal and connective tissue disorders) | 9 (14)
Dermatology / Skin - Other (Skin and subcutaneous tissue disorders) | 10 (15)
Nail Changes (Skin and subcutaneous tissue disorders) | 14 (15)
Bilirubin (hyperbilirubinemia) (Investigations) | 8 (15)
Urinary frequency / urgency (Renal and urinary disorders) | 13 (15)
Edema: limb (General disorders) | 13 (17)
Dizziness (Nervous system disorders) | 12 (19)
Neuropathy: sensory (Nervous system disorders) | 11 (19)
Insomnia (Psychiatric disorders) | 15 (20)
Anorexia (Metabolism and nutrition disorders) | 18 (22)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 17 (22)
Febrile neutropenia (fever of unknown origin without documented infection) (Blood and lymphatic system disorders) | 19 (24)
Hair Loss / Alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 26 (26)
Constipation (Gastrointestinal disorders) | 15 (26)
Rash / desquamation (Skin and subcutaneous tissue disorders) | 19 (27)
Pulmonary / Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 16 (27)
Cough (Respiratory, thoracic and mediastinal disorders) | 19 (31)
Neutrophils / granulocytes (ANC / AGC) (Investigations) | 22 (32)
Pain - Other (General disorders) | 17 (38)
Alkaline phosphatase (Investigations) | 21 (40)
Vomiting (Gastrointestinal disorders) | 25 (42)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 27 (42)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (Infections and infestations) | 27 (44)
Mucositis / Stomatitis (clinical exam) (Gastrointestinal disorders) | 28 (48)
Nausea (Gastrointestinal disorders) | 31 (49)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 32 (52)
AST, SGOT (serum glutamic oxaloacetic transaminase) (Investigations) | 30 (57)
Diarrhea (Gastrointestinal disorders) | 28 (58)
Hemoglobin (Blood and lymphatic system disorders) | 39 (96)
Platelets (Investigations) | 39 (121)
Leukocytes (total WBC) (Investigations) | 39 (139)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes